CLINICAL TRIAL: NCT06945523
Title: Clinical Study of CEA Targeting Chimeric Antigen Receptor T Lymphocytes (CAR-T) for CEA Positive Advanced Lung Cancer
Brief Title: Clinical Study on Chimeric Antigen Receptor T Lymphocyte (CAR-T) Targeting CEA for the Treatment of CEA - Positive Advanced Lung Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chongqing Precision Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PBC082
Record Dates: First submitted 2025-04-11; First posted 2025-04-25 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-04

CONDITIONS: Advanced Lung Cancer
Keywords: CEA; CAR-T; Advanced Lung Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Targeted CEA CAR-T intravenous infusion group (Experimental)
  Interventions: Biological: Targeted CEA CAR-T
- Targeting CEA CAR-T pleural infusion group (Experimental)
  Interventions: Biological: Targeted CEA CAR-T

INTERVENTIONS:
Biological: Targeted CEA CAR-T — Subjects meeting the transfusion criteria will receive pre-treatment, which is as follows: fludarabine 25mg/m2/d×3day and cyclophosphamide 300mg/m2/d×3day, and intravenous CEA CAR-T therapy after 1-2 days of rest
  Arms: Targeted CEA CAR-T intravenous infusion group
Biological: Targeted CEA CAR-T — Subjects meeting the reinfusion criteria will receive pre-treatment with fludarabine 25mg/m2/d×3day and cyclophosphamide 300mg/m2/d×3day, rest for 1-2 days, and intraperitoneal reinfusion targeted CEA CAR-T therapy
  Arms: Targeting CEA CAR-T pleural infusion group

SUMMARY:
Lung cancer is the leading cause of morbidity and mortality in the world, of which 80%-85% are non-small cell lung cancer (NSCLC). Most patients with NSCLC are at the advanced stage of diagnosis and have a poor prognosis. The 5-year survival rate of stage III patients is about 15%, the 5-year survival rate of stage IV patients is less than 5%, and the median survival time is only 7 months.

CEACAM5 (CEA), also known as CD66e, is a classic tumor marker that has been used as a marker for many types of tumors for 50 years. It is mainly expressed in lung cancer, esophageal cancer, bile duct cancer, colorectal cancer, gastric cancer and other tumor types.

In previous CAR-T-related clinical trials targeting CEA, the research team found that CAR-T cell preparations had a certain killing effect on CEA positive tumor cells. At the same time, CAR-T cell preparations cannot be sustained for a long time in the body, which is also a key factor restricting the anti-tumor effect of CAR-T cells in the body. To solve this problem, the killing ability and survival ability of CAR-T cell preparations on tumor cells in vitro and in vivo were improved by optimizing CAR structure and improving culture mode.

DETAILED DESCRIPTION:
This study is a single-arm, open, enhanced 3+3 dose-ascending + dose-extending clinical study, aiming to evaluate the safety and efficacy of CAR T cell preparations, initially observe and study the pharmacokinetic characteristics of drugs in CEA positive advanced lung cancer patients, and obtain the recommended dose of CAR T cell preparations for CEA positive advanced lung cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years, regardless of gender.
2. Histologically or cytologically confirmed diagnosis of advanced, metastatic, or recurrent lung cancer, including both non-small cell lung cancer (NSCLC) and small cell lung cancer (SCLC).
3. Disease progression or intolerance following at least one line of prior therapy (including but not limited to surgery, chemotherapy, radiotherapy, targeted therapy, or immunotherapy).
4. For patients with pleural effusion enrolled in the intrapleural infusion group, accurate assessment of pleural effusion volume and characteristics must be conducted via imaging (chest CT or X-ray) combined with cytological analysis. Cytological examination must confirm the presence of tumor cells in the pleural effusion, indicating malignant pleural effusion.
5. Positive tumor CEA expression confirmed by immunohistochemistry (IHC) within 3 months prior to screening (defined as clear membranous staining with a positivity rate ≥10%). If IHC testing of tumor samples was performed more than 3 months prior to screening, the patient's serum CEA must be >10 ng/mL.
6. At least one measurable lesion according to RECIST 1.1 criteria: for non-nodal lesions, the longest diameter must be ≥10 mm; for nodal lesions, the short axis must be ≥15 mm.
7. ECOG performance status score of 0-2.
8. Expected survival of more than 12 weeks.
9. No severe psychiatric disorders.
10. Unless otherwise specified, key organ functions must meet the following requirements:

    1. Hematologic: WBC >2.0×10⁹/L, neutrophils >1.0×10⁹/L, lymphocytes >0.5×10⁹/L, platelets >50×10⁹/L, hemoglobin >80 g/L;
    2. Cardiac function: Left ventricular ejection fraction (LVEF) ≥50% by echocardiography, and no significant abnormalities on ECG;
    3. Renal function: Serum creatinine ≤2.0×ULN;
    4. Hepatic function: ALT and AST ≤3.0×ULN (≤5.0×ULN if liver metastases are present);
    5. Total bilirubin ≤2.0×ULN;
    6. Oxygen saturation (SpO₂) >92% on room air.
11. Eligible for leukapheresis or peripheral venous blood collection and without contraindications for cell collection.
12. Subjects must agree to use reliable and effective contraception (excluding rhythm method) from the time of informed consent until 1 year after CAR-T cell infusion.
13. Subject or legally authorized representative must voluntarily sign the informed consent form (ICF), indicating understanding of the study objectives and procedures and willingness to participate in the clinical trial.

Exclusion Criteria:

1. Presence of symptomatic central nervous system (CNS) metastases or leptomeningeal metastases at screening, or other evidence indicating that CNS or leptomeningeal lesions are not adequately controlled, making the patient unsuitable for enrollment as judged by the investigator.
2. Participation in another clinical study within 1 month prior to screening.
3. Receipt of a live attenuated vaccine within 4 weeks prior to screening.
4. Prior antitumor therapies before screening including: chemotherapy, targeted therapy, or other investigational drugs administered within 14 days or at least 5 half-lives (whichever is shorter) before screening.
5. Active or uncontrolled infections requiring systemic treatment.
6. Tumor compressing the trachea or major blood vessels with high risk as assessed by the investigator.
7. Presence of any of the following cardiac conditions:

   1. New York Heart Association (NYHA) Class III or IV congestive heart failure;
   2. Myocardial infarction or coronary artery bypass graft (CABG) within 6 months prior to enrollment;
   3. Clinically significant ventricular arrhythmias or a history of unexplained syncope (excluding vasovagal or dehydration-related causes);
   4. History of severe non-ischemic cardiomyopathy.
8. Active autoimmune diseases or other conditions requiring long-term immunosuppressive therapy.
9. History of other untreated or concurrent malignancies within the past 3 years, except for adequately treated cervical carcinoma in situ or basal cell carcinoma of the skin.
10. Positive hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) with detectable hepatitis B virus (HBV) DNA levels exceeding the normal range in peripheral blood; positive hepatitis C virus (HCV) antibody with detectable HCV RNA levels exceeding the normal range in peripheral blood; positive for human immunodeficiency virus (HIV) antibodies; or positive syphilis test.
11. Pregnant or breastfeeding women.
12. Any other condition that, in the opinion of the investigator, renders the patient unsuitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-28 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of CAR T cell preparations in the treatment of CEA positive advanced lung cancer【safety】 | 28days
  Adverse events and their proportion during the trial (assessed against the Common Terminology Standard for Adverse Events Version 5.0 (CTCAE 5.0) and ASTCT standards)

SECONDARY OUTCOMES:
To evaluate the disease control rate of CAR-T cell preparations in CEA positive advanced lung cancer【efficacy】 | 3months
  Disease control rates at 3 months were assessed according to Response Evaluation Criteria in Solid Tumors,Version 1.1 (RECIST 1.1), including CR, PR, and SD
To evaluate the remission rate of CAR-T cell preparations in CEA positive advanced lung cancer【efficacy | 3months
  Objective response rates at 3 months were assessed according to RECIST 1.1, including CR, PR
To evaluate the overall survival of CAR-T cell preparations in CEA-positive advanced lung cancer【efficacy】 | 2years
  Overall survival (OS) : The time from the time the subject received CAR T cell retransfusion until death (from any cause)
To evaluate the duration of response of CAR-T cell preparations in CEA-positive advanced lung cancer【efficacy】 | 2years
  Duration of response (DOR) : the time from the first evaluation of CR, PR, or SD to the first evaluation of disease recurrence or progression or death from any cause
To evaluate the disease progression-free survival of CAR-T cell preparations in CEA-positive advanced lung cancer【efficacy】 | 2years
  Disease progression-free survival (PFS) : the time from the time the subject received CAR T cell therapy until the first disease progression or death from any cause
To obtain the cytodynamics data of CAR-T cells in vivo【pharmacokinetics】 | 3months
  Cmax:The highest concentration of CAR T cells amplified in peripheral blood after reinfusion
To obtain the cytodynamics data of CAR-T cells in vivo【pharmacokinetics】 | 3months
  Tmax:The time to reach the highest concentration of CAR-T cells in peripheral blood after reinfusion
To obtain the cytodynamics data of CAR-T cells in vivo【pharmacodynamics】 | 2years
  The content of free CEA in peripheral blood at each time point after transfusion was determined by immunohistochemical method

CONTACTS AND LOCATIONS:
Locations (1):
- Wuhan Pulmonary Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No